CLINICAL TRIAL: NCT00680264
Title: Prospective Database Registry Study of Scoliosis in Children With Cerebral Palsy
Acronym: PCPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Setting Scoliosis Straight Foundation (Other)
Collaborators: K2M, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2007HSG021
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Palsy; Scoliosis
Keywords: Treatment Outcomes; Scoliosis; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Operative: Diagnosis of Cerebral Palsy (standard definition of any brain injury before the age of 3) with total body involvement - any functional level Curve >40 degrees on sitting film, A spinal fusion is being undertaken and the patient/family is proceeding with the spinal fusion (with any level of distal fusion).
- Non-operative: Diagnosis of Cerebral Palsy (standard definition of any brain injury before the age of 3) with total body involvement - any functional level, Curve >40 degrees on sitting film, A spinal fusion is not being undertaken either because the family has refused surgery or because it is not recommended at this point.

SUMMARY:
The purpose of this study is to determine the radiographic and clinical outcomes of Scoliosis surgical and non-operative treatment in patients with Cerebral Palsy.

DETAILED DESCRIPTION:
Bracing severe neuromuscular scoliotic curves rarely serves as definitive treatment, thus most progressive curves require surgical intervention in order to sustain or improve sitting (or ambulatory) abilities. Surgery is a demanding intervention for these patients, with variable functional gains. Controversy persists regarding indications for surgery, timing, and technique. Concerns about complications are paramount. Previous neuromuscular studies have been confined to a small number of surgeons with a narrow range of surgical instrumentation, technique, and correction. Very little evidence exists regarding the impact spinal surgery on the quality of life in children with scoliosis related to cerebral palsy. The instruments to measure quality of life are not specific to children with scoliosis related to cerebral palsy. There have been no comprehensive prospective studies published. This study would be the first large-scale prospective, multi-center series of spinal fusion outcomes in patients with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 8-21 years
* Diagnosis of Cerebral Palsy (standard definition of any brain injury before the age of 3) with total body involvement - any functional level
* Coronal Curve >50 degrees on sitting film (as measured by 'greatest Cobb') OR Kyphotic curve >70 degrees on sitting film (as measured by T5-T12) AND
* A spinal fusion is being undertaken and the patient/family is proceeding with the spinal fusion (with any level of distal fusion).

OR

• A spinal fusion is not being undertaken (Non-Operative cohort) either because the family has refused surgery or because it is not recommended at this point or surgery is recommended but is not being undertaken because they are on a waiting list, and are being enrolled as a non-op patient because they will be on the waiting list for >18 months.

Exclusion Criteria:

* Previous operated scoliotic spine deformity
* Diagnosis of Rett's Syndrome
* Concomitant lower extremity surgery (within 3 months of spinal fusion)

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who present to the investigator's clinic, who meet the inclusion criteria will be offered enrollment in the study
Sampling Method: Non-Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2008-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
radiographic outcomes | 5 year

SECONDARY OUTCOMES:
Clinical outcomes | 5 years
Health related quality of life outcomes | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sponseller, MD, Principal Investigator — John's Hopkins Hospital; Peter Newton, MD, Study Director — Rady Children's Hospital San Deigo; Michelle Marks, PT, MA, Study Chair — Harms Study Group
Locations (15):
- United States (12):
  - Rady Children's Hospital, San Diego, California
  - A.I. Dupont Hospital for Children, Wilmington, Delaware
  - Miami Children's Hospital, Miami, Florida
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - New York University Hospital for Joint Diseases, New York, New York
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
  - Texas Scottish Rite Hospital, Dallas, Texas
  - Kluge Children's Rehab. Ctr., Charlottesville, Virginia
- Canada (3):
  - CHU Saint-Justine Hospital, Montreal
  - Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver

REFERENCES:
- See also: Setting Scoliosis Straight Website - highlighting the research of the Harms Study Group — http://hsg.settingscoliosisstraight.org/current-hsg-research/